CLINICAL TRIAL: NCT00770328
Title: The Effects of Pentoxifylline on PAI-1 in an Obese Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, James Muldowney, Assistant Professor, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 030497
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Plasma PAI-1 level at 0, 4, 8 weeks; Plasma hsCRP level at 0, 4, 8 weeks; Plasma TNF-a level at 0, 4, 8 weeks
MeSH Terms: conditions — Obesity | interventions — Pentoxifylline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentoxifylline (Experimental): Patients receive Pentoxifylline 400 mg po TID for 8 weeks.
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Patients take a placebo TID for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — 400mg PO TID x 8 weeks
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebo — PO TID x 8 weeks
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
PAI-1 is elevated in obese individuals. TNF-alpha, an inflammatory mediator is believed to play a role in obesity mediated elevations in PAI-1 levels. TNF-alpha blockade with antibodies and the drug pentoxifylline have been shown to lower PAI-1 levels in animal models. This study tests the hypothesis that pentoxifylline will lower PAI-1 levels in human subjects.

DETAILED DESCRIPTION:
Obese individuals with elevated PAI-1 levels (greater than 10 ng/ml) are randomized to pentoxifylline 400mg, three times a day (TID) or placebo for 8 weeks. PAI-1, TNF-a and high sensitivity C-Reactive Protein are measured at week 0, 4 and 8.

ELIGIBILITY:
Inclusions: 1. A Body Mass Index of ≥ 30.0 2. Age 21 or older 3. Few or no medical problems 4. PAI-1 level ≥ 10 ng/dl

Exclusions: 1. Cigarette use 2. Present use of angiotensin converting enzyme (ACE) Inhibitors 3. Recent cerebral and/or retinal hemorrhage 4. Intolerance to pentoxifylline or methylxanthines such as caffeine, theophylline, and theobromine 5. Presently on warfarin therapy 6. Pregnancy or breast-feeding 7. Recent surgery 8. Recent diagnosis/treatment for peptic ulcer

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-05; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A S Muldowney, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 22 | 15
Completed | 9 | 11
Not Completed | 13 | 4
Not completed — Adverse Event | 11 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 22 | 15 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Study was completed and submitted for publication in 2011. We do not have the complete data set to answer questions about patients who did not complete the study.
  years
    number analyzed (Participants) | 9 | 11 | 20
    (all) | 37.7 (3.1) | 38.6 (2.5) | 38.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study submitted for publication in 2011. Records no longer exist to answer questions about screen failures and dropouts.
  Participants
    number analyzed (Participants) | 9 | 11 | 20
    Female | 5 | 5 | 10
    Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 22 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in PAI-1 Level
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 9 | 11
ng/ml
  Baseline | 39.5 (8.3) | 31.6 (7.6)
  8 Weeks | 28.6 (7.7) | 37.9 (8.5)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in CRP Level
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 9 | 11
mg/dl
  Baseline | 5.2 (2.5) | 2.9 (0.5)
  8 weeks | 4.6 (1.9) | 2.4 (0.5)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Test type: Superiority; p = 0.0114, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in TNF-alpha Level
Time Frame: Baseline and 8 weeks
Population: TNF-a assay did not work properly. Meaningless data resulted including negative values which are impossible.
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Changes in the Relationship Between PAI-1, CRP, and TNF-a With Therapy.
Time Frame: Baseline and 8 weeks
Population: Unable to complete analysis due to TNF-a assay failure (see Outcome measure #3)
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The subjects were followed from baseline to 8 weeks.
Arm/Group | Pentoxifylline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/15
Other Adverse Events (participants affected / at risk) | 11/22 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline (N=22) | Placebo (N=15)
Nausea/Vomiting (Gastrointestinal disorders) | 11 (11) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes